CLINICAL TRIAL: NCT03461029
Title: Bispectral Index Monitoring During Anesthesiologist - Directed Sedation in Scheduled Colonoscopies
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Iratxe González Mendibil, Principal Investigator, Hospital Galdakao-Usansolo
Other Study IDs: 01/16
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Colonoscopy
Keywords: Sedation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIS: Group of 196 patients in whom sedation monitoring is performed using the Bispectral Index Monitoring (BIS) system.
  Interventions: Device: BIS monitor

INTERVENTIONS:
Device: BIS monitor — The investigators placed on the forehead of all patients the sensor BIS quatroTM, that connects with the monitor, and they registered sedation and recorded the values obtained.

SUMMARY:
The aim of the study is to establish and identify the level of sedation that is performed in the endoscopy rooms of Galdakao Hospital. To do this, the investigators used the BIS monitoring system, which obtains objective values in real time from the anesthesia performed. The monitoring is completed with basic parameters validated by European guidelines (heart rate, blood pressure, oxygen saturation and respiratory rate), capnography and Ramsay sedation scale, widely validated for use outside the operating room. The main work hypothesis was that in at least 10% of the patients BIS values compatible with moderate or deep sedation would be obtained (BIS <65).

DETAILED DESCRIPTION:
Observational study in patients undergoing scheduled colonoscopy in endoscopy rooms of the Galdakao-Usansolo Hospital. The investigators objectified the level of sedation that was performed in these procedures using Bispectral Index Monitoring, as well as the total dose of medication required and the level of satisfaction obtained after completing the sedation. The incidence of hemodynamic and respiratory complications observed was included, as well as the treatment needed to solve them.

A total of 196 patients were needed to obtain statistically significant results. Qualitative variables are expressed in the form of freguencies and percentages and continuous variables in the form of means and stnadard deviations. Comparisions of percentages were made by the Chi square test and the difference of means in the continuous variables by the t test.Stadistical significance will be assumed when p<0.05. All estadistical analyzes were carried out using SAS V9.4 (SAS Institute, Inc., Carey, NC).

ELIGIBILITY:
Inclusion Criteria:

* Indication of scheduled colonoscopy.
* Classification of physical status ASA I, II and III.
* Intermitent or persistent mild asthma.
* Body Mass Index (BMI) < 35 kg/m2.
* Intact neurological capacity.
* Acceptance to participate in the study after signing written informed consent.

Exclusion Criteria:

* ASA IV.
* BMI > 35 kg/m2.
* Allergy to any of the medications using in sedation, or its components.
* Known mental or neurological disease.
* Chronic Obstructive Pulmonary Disease (COPD) or Obstructive Sleep Apnea.
* Chronic opiate users.
* Refusal to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the general population, residents in the geographical area corresponding to the Hospital Galdakao Usansolo, who attended the endoscopy rooms. Were included to undergo a scheduled colonoscopy, either for monitoring, diagnostic or screening, and to meet the cited inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Level of sedation | 1 year.
  Sedation measured by Bispectral Index Monitoring.

SECONDARY OUTCOMES:
Complications related to sedation. | 1 year.
  Complications were measured: hypotension, bradicardia, apnea and low oxygen saturation. The medications or maneuvers that were necessary to correct these complications were also evaluated.
Level of satisfaction with the sedation. | 1 year.
  The investigators distributed a satisfaction questionnaire to all patients after colonoscopy to find their opinion about the quality of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Iratxe Gonzalez Mendibil, MD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The information contained in the study will be published once the review of the data included in it is completed. Previously, researchers will decide if the information contained is relevant for publication on this platform.

REFERENCES:
- [Background] Dumonceau JM, Riphaus A, Schreiber F, Vilmann P, Beilenhoff U, Aparicio JR, Vargo JJ, Manolaraki M, Wientjes C, Racz I, Hassan C, Paspatis G. Non-anesthesiologist administration of propofol for gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates Guideline--Updated June 2015. Endoscopy. 2015 Dec;47(12):1175-89. doi: 10.1055/s-0034-1393414. Epub 2015 Nov 12. No abstract available. PMID 26561915
- [Background] Park WY, Shin YS, Lee SK, Kim SY, Lee TK, Choi YS. Bispectral index monitoring during anesthesiologist-directed propofol and remifentanil sedation for endoscopic submucosal dissection: a prospective randomized controlled trial. Yonsei Med J. 2014 Sep;55(5):1421-9. doi: 10.3349/ymj.2014.55.5.1421. PMID 25048506
- [Background] Lera dos Santos ME, Maluf-Filho F, Chaves DM, Matuguma SE, Ide E, Luz Gde O, de Souza TF, Pessorrusso FC, de Moura EG, Sakai P. Deep sedation during gastrointestinal endoscopy: propofol-fentanyl and midazolam-fentanyl regimens. World J Gastroenterol. 2013 Jun 14;19(22):3439-46. doi: 10.3748/wjg.v19.i22.3439. PMID 23801836
- [Background] Yu YH, Han DS, Kim HS, Kim EK, Eun CS, Yoo KS, Shin WJ, Ryu S. Efficacy of bispectral index monitoring during balanced propofol sedation for colonoscopy: a prospective, randomized controlled trial. Dig Dis Sci. 2013 Dec;58(12):3576-83. doi: 10.1007/s10620-013-2833-4. Epub 2013 Aug 28. PMID 23982208
- [Background] Imagawa A, Fujiki S, Kawahara Y, Matsushita H, Ota S, Tomoda T, Morito Y, Sakakihara I, Fujimoto T, Taira A, Tsugeno H, Kawano S, Yagi S, Takenaka R. Satisfaction with bispectral index monitoring of propofol-mediated sedation during endoscopic submucosal dissection: a prospective, randomized study. Endoscopy. 2008 Nov;40(11):905-9. doi: 10.1055/s-2008-1077641. PMID 19023932
- [Background] Bower AL, Ripepi A, Dilger J, Boparai N, Brody FJ, Ponsky JL. Bispectral index monitoring of sedation during endoscopy. Gastrointest Endosc. 2000 Aug;52(2):192-6. doi: 10.1067/mge.2000.107284. PMID 10922090